CLINICAL TRIAL: NCT07139249
Title: Impact of Gender Difference and Exercise Intensities on Depression and Anxiety Symptoms Among University Students
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya Mohammed Hassan, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Aya-Phd
Record Dates: First submitted 2025-08-17; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Depression; Anxiety; University Students; Gender; Exercise Intensity
MeSH Terms: conditions — Depression; Anxiety Disorders; Coitus

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- females with high intensity interval training (Experimental): It will consist of 14 female students; they will be receiving high intensity interval training.
  Interventions: Other: The high intensity interval training
- males with high intensity interval training (Active Comparator): It will consist of 14 male students; they will be receiving high intensity interval training.
  Interventions: Other: The high intensity interval training
- females with moderate intensity continuous training. (Experimental): It will consist of 14 female students; they will be receiving moderate intensity continuous training
  Interventions: Other: The study moderate continuous training
- males with moderate intensity continuous training. (Active Comparator): It will consist of 14 male students; they will be receiving moderate intensity continuous training
  Interventions: Other: The study moderate continuous training
- The non-exercise females group (No Intervention): It will consist of 14 female students; they will remain sedentary for the six-weeks intervention period.
- The non-exercise males group (No Intervention): It will consist of 14 male students; they will remain sedentary for the six-weeks intervention period

INTERVENTIONS:
Other: The high intensity interval training — The training program for students in groups 1 and 2 involves high intensity interval training exercises, conducted three times per week for six weeks. The sessions include a 10-minute warm-up at 40% Heart Rate Reserve, four high-intensity work periods at 85-95% Heart Rate Reserve, three low-intensity work periods at 60-70% Heart Rate Reserve, and a 5- 10 minute cool down at 30% Heart Rate Reserve.
  Arms: females with high intensity interval training; males with high intensity interval training
Other: The study moderate continuous training — All students in groups 3&4 will receive moderate continuous training 3 times per week for 6 weeks. Each session 40 to 50 minutes included a 5 to 10 minute warm-up, fo followed by 30 minutes of moderate aerobic exercise (treadmill walking exercise) with constant intensity at 60% to 70% Heart Rate Reserve and 5 to 10 minutes cool-down
  Arms: females with moderate intensity continuous training.; males with moderate intensity continuous training.

SUMMARY:
This study was done to investigate the impact of gender differences and exercise intensities on depression and anxiety symptoms among university students

DETAILED DESCRIPTION:
Depression among university students is a growing concern due to factors such as separation from family, transition to a performance-based environment, financial stressors, and uncertainty about postgraduation. An estimated 71% of Egyptian university students have at least minor depression. Depression is associated with lower academic performance and can lead to substance abuse, chronic conditions, and premature mortality. Despite the availability of effective treatment, only one in five university students receives minimally adequate treatment. Physical exercise is suggested as an affordable, low-cost, non-pharmacological treatment for depression and anxiety. Exercise can effectively relieve anxiety symptoms, and a study will evaluate depression and anxiety symptoms based on gender and exercise intensity among university students.

ELIGIBILITY:
Inclusion Criteria:

* Being a student in higher education
* Being single
* Age between 18 and 25 years of both sexes
* Accepting the principle of randomization in the trial.
* The body mass index is 18.5-24.9 kg/m².
* Diagnosed by psychiatrist as having a mild to moderate degree of anxiety and depression.
* Having scores of 7-24 on the Hamilton Rating Scale for Depression.
* Having scores of 17-30 on the Hamilton Anxiety Rating Scale.

Exclusion Criteria:

* Neurological history such as illness or head trauma
* Present severe and unstable respiratory disease
* History of heart defect or cardiovascular disease or any other medical conditions prohibiting high-intensity sport or physical activity
* Being professional athlete.
* Involved in regular routine of exercises
* Taking medication for mental health history of any neurological disorders like neuropathy or seizures.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-08-20 (Estimated); Primary Completion 2026-01-20 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
assessment of the severity of depressive symptoms | at baseline and after 6 weeks
  The Hamilton Rating Scale for Depression will be used to assess the severity of depressive symptoms in students across six groups. The 17-item version ranges from 0 to 54, with scores ranging from 0 to 24. Scores between 0 and 6 indicate no depression, while scores between 7 and 17 indicate mild, 18-24 indicate moderate, and 24+ over 24 indicate severe depression. A decrease in scores of at least 50% indicates response, and scores of 7 or less after treatment indicate remission. The 17-item version has adequate reliability and validity.

SECONDARY OUTCOMES:
assessment of severity of perceived anxiety symptoms | at baseline and after 6 weeks
  The Hamilton Rating Scale for Anxiety is a tool used to assess the severity of perceived anxiety symptoms. It consists of 14 symptom-defined elements, scoring from 0 to 4 (severe). The score range is 0 to 56, with scores above 17/56 indicating mild anxiety, 25-30 indicating moderate anxiety, and >30 indicating severe anxiety. It has good psychometric properties.
assessment of physical fitness | at baseline and after 6 weeks
  The Harvard Step Test is a physical fitness index that measures an individual's ability to recover from muscular work and perform muscular tasks. It is performed on a 33 cm bench at 30 steps per minute, with heart rate measured every two seconds. The test is valid for estimating the cardiorespiratory fitness of college students and can be divided into three categories: excellent, good, average, and poor. The physical efficiency index rating ranges from 96 to 115, with the highest rating being excellent for males and the lowest being poor. The test is a reliable tool for assessing physical fitness.
assessment of heart rate during exercise | at baseline and after 6 weeks
  A pulse oximeter will be used to continuously monitor heart rate during exercise, ensuring the target heart rate (THR) remains within the pre-calculated value. The heart rate will be measured and monitored for all participants using the Karvonen formula. The process involves cleaning the index finger, placing the pulse oximeter on the index, and keeping the pulse for at least a minute until the reading stabilizes.

CONTACTS AND LOCATIONS:
Locations (1):
- out-patient clinic, faculty of physical therapy, Horus university, Damietta, Egypt